CLINICAL TRIAL: NCT05204758
Title: Prophylactic TCM for Mitigation of EGFR-TKI Related Dermatological Adverse Effect
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMUH105-REC1-055
Record Dates: First submitted 2021-12-23; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Advanced Lung Adenocarcinoma
Keywords: advanced lung adenocarcinoma; EGFR-TKI; traditional Chinese medicine; skin toxicity; quality of life; prophylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Experimental): Patients receive afatinib and TCM. TCM recipe was chosen from three essential TCM formulas, including Bai He Gu Jin Tang (yin nourishing), Wen Dan Tang (phlegm reducing), and Qing Shang Fang Fen Tang (heat clearing). The packages contained 1.6 g TCM preparations, which were manufactured in powder form by Sun Ten Pharmaceutical (Taichung, Taiwan) according to the good manufacturing practice requirements. Patients were instructed to intake three packages of TCM preparations with each meal three times a day, for a total of nine packages per day. Administration of TCM was initiated at the same time as afatinib and continued for a total of three months.
  Interventions: Drug: TCM Formula
- Control arm (Placebo Comparator): Patients receive afatinib and placebo. Placebo without the medical ingredients was prepared to be similar to the weight, color, smell, taste, and packaging of the TCM formulas. The packages contained 1.6 g placebo preparations, which were manufactured in powder form by Sun Ten Pharmaceutical (Taichung, Taiwan) according to the good manufacturing practice requirements. Patients were instructed to intake three packages of placebo preparations with each meal three times a day, for a total of nine packages per day. Administration of placebo was initiated at the same time as afatinib and continued for a total of three months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TCM Formula — three packages of TCM preparations with each meal three times a day
  Arms: Study arm
Drug: Placebo — three packages of placebo preparations with each meal three times a day
  Arms: Control arm

SUMMARY:
Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) have become standard practice for advanced non-small cell lung cancer (NSCLC) with EGFR gene mutation. EGFR-TKIs involving Afatinib, Erlotinib, and Gefitinib were Food and Drug Administration (FDA) approved since 2006 and given payment continuously for lung adenocarcinoma with EGFR mutation in Taiwan.

Several researches mention the positive correlation between skin toxicities and clinical response, such as improved median survival, overall survival and progression-free survival. Nevertheless, quite a few patients reduced dose or discontinued EGFR-TKIs because of prolonged or intolerable adverse effects, thus causing disease progress and even death. Based on the experts' opinion, some basic strategies have been developed to manage dermatologic adverse effects. Those strategies have the potential to improve patient quality of life and to prevent dose reductions or discontinuation.

The concept of prophylaxis in EGFR-TKI related adverse effects had existed for rash and diarrhea, but it is not well spread. Although several studies indicate that Traditional Chinese Medicine (TCM) facilitates the treatment of lung cancer, clinical analysis of prophylactic TCM in EGFR-TKIs related skin toxicities remains absent. Based on TCM syndrome differentiation and treatment and clinical experiences, the investigators have found effective TCM compositions to relieve these toxicities.

Therefore, the investigators develop a pilot, prospective, double-blinded, randomized controlled TCM research to prevent EGFR- TKIs related dermatological adverse effects. The purpose of this study suggest that TCM could provide synergic effect with EGFR-TKIs, which means TCM could reduce and prevent EGFR-TKIs related dermatological adverse effects without interfering formulary cancer therapy. The investigators hypothesize that prophylactic TCM with standard of care will delay any grade skin toxicity to 14 days as well as reduce the incidence of grade 3 skin toxicity from 30% to less than 10%.

Due to high EGFR mutation rate of lung adenocarcinoma in Taiwan, it is necessary to investigate whether combination of TCM is beneficial to patients of advanced lung adenocarcinoma with EGFR gene mutation.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths worldwide. According to National Comprehensive Cancer Network (NCCN) Guidelines, EGFR-TKIs have become standard practice for advanced NSCLC with EGFR gene mutation. An epidemiological study in 2012 reported that EGFR mutations from Asian advanced lung adenocarcinoma patients were 22-64% and the rate in Taiwan was 62.1%. Another epidemiological study in 2015 showed that the EGFR mutation rate of treatment -naïve lung adenocarcinoma in Taiwan was 55.4%.

Depend on several extensive studies, oral treatment of EGFR-TKIs improved progression free survival (PFS) about 9.2-13.6% than traditional chemotherapy. EGFR-TKIs involving Afatinib, Erlotinib, and Gefitinib were FDA approved since 2006 and given payment continuously for lung adenocarcinoma with EGFR mutation in Taiwan.

Several researches mention the positive correlation between skin toxicities and clinical response, such as improved median survival, overall survival and progression-free survival. Nevertheless, quite a few patients reduced dose or discontinued EGFR-TKIs because of prolonged or intolerable adverse effects, thus causing disease progress and even death. Based on the experts' opinion, some basic strategies have been developed to manage dermatologic adverse effects. Those strategies have the potential to improve patient quality of life and to prevent dose reductions or discontinuation.

The concept of prophylaxis in EGFR-TKI related adverse effects had existed for rash and diarrhea, but it is not well spread. Although several studies indicate that TCM facilitates the treatment of lung cancer, clinical analysis of prophylactic TCM in EGFR-TKIs related skin toxicities remains absent. Based on TCM syndrome differentiation and treatment and clinical experiences, the investigators have found effective TCM compositions to relieve these toxicities.

Therefore, the investigators develop a pilot, prospective, double-blinded, randomized controlled TCM research to prevent EGFR- TKIs related dermatological adverse effects. The purpose of this study suggest that TCM could provide synergic effect with EGFR-TKIs, which means TCM could reduce and prevent EGFR-TKIs related dermatological adverse effects without interfering formulary cancer therapy. The investigators hypothesize that prophylactic TCM with standard of care will delay any grade skin toxicity to 14 days as well as reduce the incidence of grade 3 skin toxicity from 30% to less than 10%.

Due to high EGFR mutation rate of lung adenocarcinoma in Taiwan, it is necessary to investigate whether combination of TCM is beneficial to patients of advanced lung adenocarcinoma with EGFR gene mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of locally advanced or metastatic lung adenocarcinoma with EGFR mutations,
2. Patients with an Eastern Cooperative Oncology Group performance status score of 0-2,
3. Patients receiving afatinib as first-line treatment to ensure a shorter time to observe skin adverse effects of any grade,
4. Patients with measurable disease evaluated by the Response Evaluation Criteria in Solid Tumors (version 1.1),
5. Patients with brain metastases were included after adequate treatment.

Exclusion Criteria: -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
time to skin toxicity of any grade | 3 month
  Patients were instructed to maintain a diary to record the date on which skin toxicity of any grade first presented.
incidence of grade 3 skin toxicity | 3 months
  Patients were instructed to maintain a diary to record the date on which maximum EGFR-TKI-related skin toxicities occurred.

SECONDARY OUTCOMES:
safety evaluation | 3 months
  Safety evaluation included complete blood and differential counts, renal and liver function tests, and tumor markers.
quality of life evaluation | 3 months
  Quality of life evaluation included Dermatology Life Quality Index, Functional Assessment of Cancer Therapy-Lung (FACT-L; version 4), European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer (EORTC QLQ-C30/LC13 version 3.0), and Eastern Cooperative Oncology Group performance status (ECOG PS) scale.
progression free survival | 3 years
  Tumor response to EGFR-TKIs was assessed by chest X-ray once a month and chest computed tomography once every three months.
overall survival | 3 years
  Tumor response to EGFR-TKIs was assessed by chest X-ray once a month and chest computed tomography once every three months.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsiang Li, Attending, Principal Investigator — China Medical University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melosky B, Leighl NB, Rothenstein J, Sangha R, Stewart D, Papp K. Management of egfr tki-induced dermatologic adverse events. Curr Oncol. 2015 Apr;22(2):123-32. doi: 10.3747/co.22.2430. PMID 25908911
- [Background] Takeda M, Okamoto I, Nakagawa K. Pooled safety analysis of EGFR-TKI treatment for EGFR mutation-positive non-small cell lung cancer. Lung Cancer. 2015 Apr;88(1):74-9. doi: 10.1016/j.lungcan.2015.01.026. Epub 2015 Feb 7. PMID 25704957
- [Background] Melosky B, Anderson H, Burkes RL, Chu Q, Hao D, Ho V, Ho C, Lam W, Lee CW, Leighl NB, Murray N, Sun S, Winston R, Laskin JJ. Pan Canadian Rash Trial: A Randomized Phase III Trial Evaluating the Impact of a Prophylactic Skin Treatment Regimen on Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor-Induced Skin Toxicities in Patients With Metastatic Lung Cancer. J Clin Oncol. 2016 Mar 10;34(8):810-5. doi: 10.1200/JCO.2015.62.3918. Epub 2015 Nov 16. PMID 26573073
- [Background] Yang XB, Wu WY, Long SQ, Deng H, Pan ZQ. Effect of gefitinib plus Chinese herbal medicine (CHM) in patients with advanced non-small-cell lung cancer: a retrospective case-control study. Complement Ther Med. 2014 Dec;22(6):1010-8. doi: 10.1016/j.ctim.2014.10.001. Epub 2014 Oct 12. PMID 25453521
- [Background] Liu ZL, Zhu WR, Zhou WC, Ying HF, Zheng L, Guo YB, Chen JX, Shen XH. Traditional Chinese medicinal herbs combined with epidermal growth factor receptor tyrosine kinase inhibitor for advanced non-small cell lung cancer: a systematic review and meta-analysis. J Integr Med. 2014 Jul;12(4):346-58. doi: 10.1016/S2095-4964(14)60034-0. PMID 25074884
- [Derived] Li CL, Hsia TC, Yang ST, Chao KC, Tu CY, Chen HJ, Li CH. Efficacy of Prophylactic Traditional Chinese Medicine on Skin Toxicity of Afatinib in EGFR Mutation-Positive Advanced Lung Adenocarcinoma: A Single-Center, Prospective, Double-Blinded, Randomized-Controlled Pilot Trial. Integr Cancer Ther. 2022 Jan-Dec;21:15347354221086663. doi: 10.1177/15347354221086663. PMID 35297709
- See also: Management of egfr tki-induced dermatologic adverse events. — https://pubmed.ncbi.nlm.nih.gov/25908911/
- See also: Pooled safety analysis of EGFR-TKI treatment for EGFR mutation-positive non-small cell lung cancer — https://pubmed.ncbi.nlm.nih.gov/25704957/
- See also: Pan Canadian Rash Trial: A Randomized Phase III Trial Evaluating the Impact of a Prophylactic Skin Treatment Regimen on Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor-Induced Skin Toxicities in Patients With Metastatic Lung Cancer — https://pubmed.ncbi.nlm.nih.gov/26573073/
- See also: Effect of gefitinib plus Chinese herbal medicine (CHM) in patients with advanced non-small-cell lung cancer: a retrospective case-control study — https://pubmed.ncbi.nlm.nih.gov/25453521/
- See also: Traditional Chinese medicinal herbs combined with epidermal growth factor receptor tyrosine kinase inhibitor for advanced non-small cell lung cancer: a systematic review and meta-analysis — https://pubmed.ncbi.nlm.nih.gov/25074884/